CLINICAL TRIAL: NCT03022838
Title: The Effects of Caffeine Withdrawal on Migraine - a Randomized, Double-blind, Crossover Study
Brief Title: The Effects of Caffeine Withdrawal on Migraine
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The study was terminated prematurely due to poor recruitment.
Sponsor: Nordlandssykehuset HF (Other)
Collaborators: King's College London (Other); University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2015/1729REK
Record Dates: First submitted 2016-12-29; First posted 2017-01-18 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Migraine; Caffeine Withdrawal
MeSH Terms: conditions — Migraine Disorders | interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caffeine (Active Comparator): Caffeine tablets (Recip) 100 mg, 300-800 mg
  Interventions: Drug: Caffeine
- Placebo (Placebo Comparator): Placebo tablets
  Interventions: Drug: Caffeine

INTERVENTIONS:
Drug: Caffeine — From the point of enrollment, patients will substitute their daily dietary caffeine with either placebo- or capsulated caffeine tablets (Recip®, 100mg).
  Other Names: Recip

SUMMARY:
Sporadic and chronic dietary consumption of caffeine has substantial biological effects on the nervous system. The effects on migraine are at large not known. In this study we want to assess the effects of caffeine withdrawal on migraine.

DETAILED DESCRIPTION:
The actions of caffeine as an antagonist of adenosine receptors have been extensively studied, and there is no doubt that both daily and sporadic dietary consumption of caffeine has substantial biological effects on the nervous system. The current opinion is that caffeine both can cure and trigger headaches. Caffeine is a component of many combination drugs marketed for the relief of headaches, but on the other hand it is strongly incriminated as a risk factor for developing chronic headache. Withdrawal may cause symptom constellations similar to the migraine syndrome. Further, caffeine consumption may affect sleep and alertness, possibly influencing the risk of migraine attacks. .

ELIGIBILITY:
Inclusion Criteria:

* migraine present for at least 1 year and fulfilling diagnostic criteria (ICHD-3 beta)
* =/> 3 migraine attacks per month
* no migraine prophylaxis the last month
* consumption =/> 300 mg and </= 800 mg caffeine per day the last month
* signed consent

Exclusion Criteria:

* suspicion of medication-overuse headache
* pregnancy and breast feeding
* serious co-morbidity or conditions requiring Medical treatment or caution
* working night shift
* use of drugs with moderate or major interactions with caffeine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
Migraine days | 10 weeks
  Reduction from baseline in monthly migraine days (withdrawal vs. caffeine)

SECONDARY OUTCOMES:
Withdrawal symptoms and/or syndrome (according to criteria) | 2 first days after caffeine withdrawal(withdrawal vs. caffeine)
  If patients report withdrawal symptoms, these will be recorded and eventually diagnosed as either caffeine withdrawal symptoms or migraineous symptoms in accordance with international criteria
Migraine attacks | 10 weeks
  Reduction from baseline in monthly migraine attacks (withdrawal vs. caffeine)
Sleep improvement | 10 weeks
  Reduction from baseline in PSQI and measured by actigraphy (withdrawal vs. caffeine)
Quality of life | 10 weeks
  Reduction from baseline in HIT-6 (withdrawal vs. caffeine)

CONTACTS AND LOCATIONS:
Overall Officials: Jan T Henriksen, Study Director — Department for research and patient safety, Nordland Hospital trust
Locations (3):
- Norway (3):
  - Nordland Hospital, Bodø
  - Departement of Neurology, NLSH HF, Bodø
  - Departement of Neurology, Tromsø

IPD SHARING:
Plan to Share IPD: No